CLINICAL TRIAL: NCT04838912
Title: Testing a Cognitive Behavioural Therapy Program for Anxiety in Teenagers on the Autism Spectrum: A Feasibility Study
Brief Title: Testing a CBT Program for Anxiety in Teenagers With Autism: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-16-02-37-21
Record Dates: First submitted 2021-03-25; First posted 2021-04-09 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2022-11

CONDITIONS: Anxiety; Autism
Keywords: CBT; Anxiety; Autism; Feasibility; Teenagers
MeSH Terms: conditions — Anxiety Disorders; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Fifteen teenagers aged 13-17 years with an active ASD diagnosis and experiencing life interference anxiety symptoms will be divided into 3 groups and treated with the Cool Kids AST anxiety program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cool Kids ASA (Experimental): The Cool Kids (Chilled) ASA anxiety program
  Interventions: Behavioral: Cool Kids (Chilled) Anxiety program adapted to children and youths with autism and anxiety disorders.

INTERVENTIONS:
Behavioral: Cool Kids (Chilled) Anxiety program adapted to children and youths with autism and anxiety disorders. — CBT program for anxiety in teenagers with autism

SUMMARY:
The objective is to investigate the feasibility of a newly developed manualised group Cognitive Behavioural Therapy (CBT) programme for anxiety in 15 teenagers (aged 13-17 years) with Autism Spectrum Disorder (ASD). Our aim is to focus primarily on acceptability and compliance with the program with some investigation of treatment effects on anxiety diagnosis and anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Fulfil the diagnostic criteria for one or more anxiety diagnoses on the Anxiety Disorders Interview Schedule for DSM-IV: Parent & Child interview schedule (ADIS C/P)
* Obtained a diagnosis of ASD according to the International Classification of Diseases, 10th edition (ICD 10)

Exclusion Criteria:

* low intellectual functioning (<70)
* active psychosis
* untreated hyperkinetic disorder
* inability to speak Danish
* inability to leave the home
* inability to attend a group setting
* inability to meet for treatment caused by other psychiatric disorders.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
The Experience of Service Questionnaire | Interview at 14 weeks after start of treatment
  A questionnaire measuring teenagers and parents satisfaction with the treatment. On a Likert scale they will be asked to rate positive statements as 'not true' (1), 'partly true' (2), or 'true' (3) and in an open section freely comment on their experience with the treatment.

SECONDARY OUTCOMES:
Anxiety Disorders Interview Schedule for DSM-IV: Parent & Child interview schedule (ADIS C/P) | Change from baseline interview results at 14 weeks
  ADIS/CP is a structured interview involving both child and parents designed to assess for current episodes of anxiety disorders, and to permit differential diagnosis among the anxiety disorders according to DSM-IV criteria
Anxiety Disorders Interview Schedule for DSM-IV: Parent & Child interview schedule (ADIS C/P) | Change from baseline interview results at 3 months
  ADIS/CP is a structured interview involving both child and parents designed to assess for current episodes of anxiety disorders, and to permit differential diagnosis among the anxiety disorders according to DSM-IV criteria.
  With the interview the disorders are rated with a clinical severity rating (CSR) from 0 (no interference) to 8 (extreme interference) with severity ratings of 4 or above signifying the presence of a clinical disorder.
Spence Children's Anxiety Scale (SCAS) | Change from baseline results at 14 weeks
  SCAS is a questionnaire for children and parents assessing the severity of anxiety symptoms broadly in line with the dimensions of anxiety disorder proposed by the DSM-IV. The scale assesses six domains of anxiety including generalized anxiety, panic/agoraphobia, social phobia, separation anxiety, obsessive-compulsive disorder and physical injury fears.
  The items are rated on a 4 point scale: 'never','sometimes', 'often', or 'always' to indicate how often each of the items happens. A higher score means worsen of the symptom. Youth version: Min. score 0, max score 135. Parent version: Min. score 0, max score 117
Spence Children's Anxiety Scale (SCAS) | Change from baseline results at 3 months
  SCAS is a questionnaire for children and parents assessing the severity of anxiety symptoms broadly in line with the dimensions of anxiety disorder proposed by the DSM-IV. The scale assesses six domains of anxiety including generalized anxiety, panic/agoraphobia, social phobia, separation anxiety, obsessive-compulsive disorder and physical injury fears.
  The items are rated on a 4 point scale: 'never','sometimes', 'often', or 'always' to indicate how often each of the items happens. A higher score means worsen of the symptom. Youth version: Min. score 0, max score 135. Parent version: Min. score 0, max score 117
Children's Anxiety Life Inference Scale (CALIS) | Change from baseline results at 14 weeks
  CALIS is designed to assess life interference attributed to fears and worries from child and parent perspectives. The measure targets interference on the child's life and on the parent's/family's life.
  The items are rated on a 5 point scale: 'not at all', 'only a little','sometimes', 'quite a lot', or 'a great deal' to indicate how much impact each of the items has on daily life. A higher score means worsen of the impact. Youth version: Min. score 0, max score 9. Parent version: Min. score 0, max score 64
Children's Anxiety Life Inference Scale (CALIS) | Change from baseline results at 3 months
  CALIS is designed to assess life interference attributed to fears and worries from child and parent perspectives. The measure targets interference on the child's life and on the parent's/family's life.
  The items are rated on a 5 point scale: 'not at all', 'only a little','sometimes', 'quite a lot', or 'a great deal' to indicate how much impact each of the items has on daily life. A higher score means worsen of the impact. Youth version: Min. score 0, max score 9. Parent version: Min. score 0, max score 64
Children's Automatic Thoughts Scale (CATS) | Change from baseline results at 14 weeks]
  CATS is a developmentally sensitive, general measure of negative self-statements across both internalizing and externalizing problems. Four separate subscales of cognitive content are assessed including physical threat, social threat, personal failure, and hostility.
  The items are rated on a 5 point scale: 'not at all','sometimes', 'quite often', 'often' or 'all the time' to indicate how often each of the items occurs. A higher score means increase of the event. Min. score 0, max score 160.
Children's Automatic Thoughts Scale (CATS) | Change from baseline results at 3 months
  CATS is a developmentally sensitive, general measure of negative self-statements across both internalizing and externalizing problems. Four separate subscales of cognitive content are assessed including physical threat, social threat, personal failure, and hostility.
  The items are rated on a 5 point scale: 'not at all','sometimes', 'quite often', 'often' or 'all the time' to indicate how often each of the items occurs. A higher score means increase of the event. Min. score 0, max score 160.

CONTACTS AND LOCATIONS:
Locations (1):
- Auhus University Hospital, Psychiatry, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared. Only overall data on the group will be shared due to the Danish Data Protection Act.

DOCUMENTS (1):
  • Study Protocol (2021-04-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT04838912/Prot_001.pdf